CLINICAL TRIAL: NCT02287181
Title: A Phase IV Study to Investigate the Effects of Varied Remifentanil Concentrations on Propofol Requirements for Loss of Consciousness, Response to Painful Stimuli, Bispectral Index and Associated Haemodynamic Changes
Brief Title: A Phase IV Study Investigating the Effects of Remifentanil Concentrations on Propofol Requirements for Loss of Consciousness, Response to Painful Stimuli, Bispectral Index and Associated Haemodynamic Changes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Hannah Scott, Clinical Associate, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: uhongkong
Record Dates: First submitted 2014-10-24; First posted 2014-11-10 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Induction of Anaesthesia
MeSH Terms: interventions — Remifentanil; Propofol; Consciousness Monitors

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- remifentanil effect site concentration 0ng/ml (Active Comparator): remifentanil run as an infusion using the minto TCI model, at an effect site concentration of 0 nano grams per millilitre, commenced from start of proposal infusion to point at which patient is anaesthetised and not responding to painful stimuli.
  Interventions: Drug: Remifentanil; Drug: Propofol; Other: Bispectral index
- remifentanil effect site concentration 3ng/ml (Active Comparator): remifentanil run as an infusion using the minto TCI model, at an effect site concentration of 3 nano grams per millilitre, commenced from start of proposal infusion to point at which patient is anaesthetised and not responding to painful stimuli.
  Interventions: Drug: Remifentanil; Drug: Propofol; Other: Bispectral index

INTERVENTIONS:
Drug: Remifentanil — short acting opiate
Drug: Propofol — hypnotic drug
Other: Bispectral index — electroencephalograph

SUMMARY:
A prospective, randomised, phase IV trial including 150 patients.

To evaluate the effects of varied concentrations of remifentanil on the proposal requirements for the loss of consciousness and response to pain and to evaluate the haemodynamic changes and processed EEG (BIS) during induction of anaesthesia.

DETAILED DESCRIPTION:
BackGround

The combination of remifentanil and propofol infusions is a widely used method of total intravenous anaesthesia. (1) Target controlled infusion (TCI) is a pharmacokinetic (PK) infusion system using data from a large population of patients to calculate and deliver stable concentrations of a drug based on a three compartment PK model. Both propofol and remifentanil are ideal drugs for delivery in this way because of their quick distribution, metabolism and excretion. (2) Remifentanil is a potent synthetic opioid receptor (MOR) agonist with a short recovery irrespective of the duration of its administration. This is due to it being quickly broken down by non-specific esterases in blood and tissues. (3) Remifentanil like all opioids is not very hypnotic in clinically relevant concentrations. (4)

Remifentanil has been shown to reduce propofol requirements during induction and maintenance of anaesthesia. (5)(6) Also modest doses of remifentanil markedly reduce the amount of propofol required to ablate response to painful stimuli. The relationship between propofol and remifentanil has been reported as synergistic but additive when using propofol concentrations within the clinical range. (7)(8) However in other studies, BIS has shown no interaction between propofol and remifentanil (9)(10) A correlation between BIS, painful stimuli and other opioids has been demonstrated. (11) It has been suggested that BIS values can change with propofol and painful stimuli and this can aid administration of remifentanil in a dose dependent manner. (12) Since propofol and remifentanil are ubiquitously used together, the interaction between these drugs and EEG needs to be defined in more detail.

Trial Objectives To see whether remifentanil affects the dose of proposal required for loss of consciousness and loss of response to painful stimuli and whether this is reflected in changes in brain EEG (bispectral index BIS)

Hypothesis That the effect site concentration of proposal at loss of consciousness will only be moderately affected by concurrently remifentanil infusion but BIS will not change. That the clinical response to painful stimuli will markedly decrease when there is concurrent infusion of remifentanil. With painful stimuli there will be an increase in BIS but this will be blocked by remifentanil.

Methodology From the start date of the study, the first 100 patients eligible will be included. Patients will be allocated into one of two groups, group A or group B by a computer generated randomization table.

For each patient, after receiving written consent, the patient will enter the theatre where they are going to have their elective operation. Standard anaesthetic monitoring will be applied, plus a BIS monitor. External peripheral nerve stimuli electrodes will be placed over the ulner nerve on the dominant arm. IV access will be gained by the anaesthetist. All infusions will run through the same IV cannula using standardized one way valves.

One anaesthetist will look after the air way while the second anesthetist or a research assistant will fill in the data collection sheet and determine point of loss of consciousness and point of loss of response to painful stimuli. The air way anesthetist will know by a sealed envelope whether the patient is on group A or B. For the patients in group A, the remifentanil infusion, using the minto effect site concentration model, will be set at 0ng/ml. For the patients in group B the remifentanil infusion will be set at 3ng/ml. After 5 minutes the propofol infusion will commence, using the Marsh effect site concerntration TCI model, at 1mcg/ml and will be increased by 0.2mcg/ml every one minute. Heart Rate, blood pressure and BIS number will be recorded every minute. Every 30 seconds the anaesthetist will prompt the patient with the vocal stimuli "say your name" in a constant tone and volume. Loss of consciousness will be defined as the point at which the patient fails to respond to the vocal stimuli and light tactite stilulation. At this point BIS, heart rate, blood pressure and propofol effect site concentration will be recorded.

After loss of consciousness, a tetanic stimuli will be applied using the peripheral nerve stimulator and repeated every thirty seconds. The propofol infusion will continue to be increased every one minutes by 0.2mcg/ml. Loss of response to painful stimuli will be defined as the point at which the patient fails to make a withdrawal motion from the tetanic stimulation. Here, heart rate, blood pressure BIS number and propofol effect site concentration will be recorded.

After loss of response to painful stimuli the study is complete, no further date will be collected, the peripheral nerve stimulator will be removed, the anaesthesia will continue and surgery will commence as usual.

ELIGIBILITY:
Inclusion Criteria:

ASA I or II patients (healthy or with mild systemic illness) undergoing planned surgery requiring general anaesthetic

Exclusion Criteria:

1. Subjects with pre-existing neurological or psychiatric illness.
2. Subjects on CNS acting medication or analgesics.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Effect site concentration of propofol at time of loss of consciousness for each of the two groups | every 1 minute up to 40 minutes
Effect site concentration of propofol at loss of response to painful stimuli for each of the three groups | every 1 minute up to 40 minutes

SECONDARY OUTCOMES:
Time to loss of consciousness | every 1 minute up to 40 minutes
EEG Bispectral index BIS | every 1 minute up to 40 minutes
heart rate | every 1 minute up to 40 minutes
blood pressure | every 1 minute up to 40 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Michael Irwin, MbChB, Study Chair — Hong Kong University
Locations (1):
- Queen Mary Hospital, Pok Fu Lam, Hong Kong

REFERENCES:
- [Background] Vuyk J, Mertens MJ, Olofsen E, Burm AG, Bovill JG. Propofol anesthesia and rational opioid selection: determination of optimal EC50-EC95 propofol-opioid concentrations that assure adequate anesthesia and a rapid return of consciousness. Anesthesiology. 1997 Dec;87(6):1549-62. doi: 10.1097/00000542-199712000-00033. No abstract available. PMID 9416739
- [Background] Absalom AR, Mani V, De Smet T, Struys MM. Pharmacokinetic models for propofol--defining and illuminating the devil in the detail. Br J Anaesth. 2009 Jul;103(1):26-37. doi: 10.1093/bja/aep143. Epub 2009 Jun 10. PMID 19520702
- [Background] Minto CF, Schnider TW, Egan TD, Youngs E, Lemmens HJ, Gambus PL, Billard V, Hoke JF, Moore KH, Hermann DJ, Muir KT, Mandema JW, Shafer SL. Influence of age and gender on the pharmacokinetics and pharmacodynamics of remifentanil. I. Model development. Anesthesiology. 1997 Jan;86(1):10-23. doi: 10.1097/00000542-199701000-00004. PMID 9009935
- [Background] Iselin-Chaves IA, Flaishon R, Sebel PS, Howell S, Gan TJ, Sigl J, Ginsberg B, Glass PS. The effect of the interaction of propofol and alfentanil on recall, loss of consciousness, and the Bispectral Index. Anesth Analg. 1998 Oct;87(4):949-55. doi: 10.1097/00000539-199810000-00038. PMID 9768800
- [Background] Mertens MJ, Olofsen E, Engbers FH, Burm AG, Bovill JG, Vuyk J. Propofol reduces perioperative remifentanil requirements in a synergistic manner: response surface modeling of perioperative remifentanil-propofol interactions. Anesthesiology. 2003 Aug;99(2):347-59. doi: 10.1097/00000542-200308000-00016. PMID 12883407
- [Background] Jee YS, Hong JY. Effects of remifentanil on propofol requirements for loss of consciousness in target-controlled infusion. Minerva Anestesiol. 2008 Jan-Feb;74(1-2):17-22. PMID 18216764
- [Background] Bouillon TW, Bruhn J, Radulescu L, Andresen C, Shafer TJ, Cohane C, Shafer SL. Pharmacodynamic interaction between propofol and remifentanil regarding hypnosis, tolerance of laryngoscopy, bispectral index, and electroencephalographic approximate entropy. Anesthesiology. 2004 Jun;100(6):1353-72. doi: 10.1097/00000542-200406000-00006. PMID 15166553
- [Background] Ropcke H, Konen-Bergmann M, Cuhls M, Bouillon T, Hoeft A. Propofol and remifentanil pharmacodynamic interaction during orthopedic surgical procedures as measured by effects on bispectral index. J Clin Anesth. 2001 May;13(3):198-207. doi: 10.1016/s0952-8180(01)00255-0. PMID 11377158
- [Background] Guignard B, Menigaux C, Dupont X, Fletcher D, Chauvin M. The effect of remifentanil on the bispectral index change and hemodynamic responses after orotracheal intubation. Anesth Analg. 2000 Jan;90(1):161-7. doi: 10.1097/00000539-200001000-00034. PMID 10624998
- [Background] Lysakowski C, Dumont L, Pellegrini M, Clergue F, Tassonyi E. Effects of fentanyl, alfentanil, remifentanil and sufentanil on loss of consciousness and bispectral index during propofol induction of anaesthesia. Br J Anaesth. 2001 Apr;86(4):523-7. doi: 10.1093/bja/86.4.523. PMID 11573626
- [Background] Liu N, Chazot T, Hamada S, Landais A, Boichut N, Dussaussoy C, Trillat B, Beydon L, Samain E, Sessler DI, Fischler M. Closed-loop coadministration of propofol and remifentanil guided by bispectral index: a randomized multicenter study. Anesth Analg. 2011 Mar;112(3):546-57. doi: 10.1213/ANE.0b013e318205680b. Epub 2011 Jan 13. PMID 21233500